CLINICAL TRIAL: NCT06278389
Title: Study of Single Ascending Dose, Food Effects and Drug-Drug Interactions of ACC017 Tablets in Healthy Adult Participants in China: A Single-center, Randomized, Double-blind, Placebo-controlled, Two-Stage Trial
Brief Title: Single Ascending Dose, Food Effects and Drug-Drug Interactions of ACC017 Tablets in Healthy Adult Participants
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu Aidea Pharmaceutical Group Co., Ltd. (Industry)
Collaborators: Chengdu Aidea Pharmaceutical Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: ADYY-ACC017-101; CTR20240167 (Registry Identifier: chinadrugtrials.org.cn)
Record Dates: First submitted 2024-01-23; First posted 2024-02-26 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-01

CONDITIONS: Healthy Adult Participants
MeSH Terms: interventions — Emtricitabine; emtricitabine tenofovir alafenamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stage 1: ACC017 and placebo (Experimental): The trial is conducted sequentially from the low-dose cohorts, namely, 5 mg, 20 mg, 40 mg, 80 mg, 120 mg and 160 mg（tentative), respectively. Participants are given a single dose of ACC017 tablets or placebo under the fasting condition.
  Interventions: Drug: ACC017 tablets
- Stage 2: ACC017 and FTC/TAF (Descovy） (Experimental): Stage 2 is a single center, randomized, open-label FE and DDI study with a tentative dose of 40 mg. The stage was planned to enroll 12 healthy participants (both male and female) who are randomly assigned to either the fasting-postprandial or postprandial-fasting arm at a 1:1 ratio. Eligible healthy participants are admitted on D-1 and received a single oral dose of ACC017 tablets on the day of administration of each cycle under the fasting or postprandial condition with a washout period of 7 days during the two-week period. After completing the washout of the second cycle, participants are assessed by the investigator to enter into the DDI study and receive a single oral dose of ACC017 tablets with FTC/TAF tablets under the fasting condition.
  Interventions: Drug: ACC017 tablets; Drug: Emtricitabine and Tenofovir Alafenamide Fumarate Tablets

INTERVENTIONS:
Drug: ACC017 tablets — ACC017 tablets 5 mg, 20 mg, 40 mg, 80 mg, 120 mg, and 160 mg (tentative) with matching placebo
  Other Names: ACC017/Placebo
Drug: Emtricitabine and Tenofovir Alafenamide Fumarate Tablets — Participants received a single oral dose of ACC017 tablets with emtricitabine and tenofovir alafenamide fumarate tablets under the fasting condition.
  Other Names: Descovy
  Arms: Stage 2: ACC017 and FTC/TAF (Descovy）

SUMMARY:
The objective of this clinical trial is to investigate the safety and tolerability of single ascending dose ACC017 tablets in Chinese healthy adult participants. This study aims to address the following major questions:

* Recommended dosage for ACC017 tablets used in phase Ib/IIa trial;
* The pharmacokinetic (PK) characteristics of single dose ACC017 tablets;
* The effect of food (FE) on the PK of ACC017 tablets;
* Drug-drug interactions (DDIs) when ACC017 tablets are co-administered with emtricitabine and tenofovir alafenamide fumarate (FTC/TAF) tablets (II).

DETAILED DESCRIPTION:
This is a single-center, randomized, double-blind, placebo-controlled, single ascending dose (SAD), two-stage, phase Ia clinical trial in Chinese healthy adults to evaluate the safety, tolerability, PK, FE, and DDIs with FTC/TAF of ACC017 tablets administered as a single dose in healthy participants.

The trial will be divided into two stages: the first stage is a single-center, randomized, double-blind, placebo-controlled SAD study. The study consists of six dose cohorts, namely, 5 mg, 20 mg, 40 mg, 80 mg, 120 mg, and 160 mg cohorts (whether to escalate to the 160 mg cohort will be determined or adjusted if applicable) (D2~D7), and a subsequent discharge visit (D8). Participants will receive a single oral dose of ACC017 tablets or placebo under fasting conditions.

The second stage is a single-center, randomized, open-label FE and DDI study with a tentative dose of 40 mg. The final administered dose will be determined after completion of the SAD study, as assessed by the investigator and the sponsor. Stage 2 is planned to enroll 12 healthy participants (both males and females), who are randomly assigned at a 1:1 ratio to either the fasting-postprandial group (F-P group) or the postprandial-fasting group (P-F group), with 6 participants in each group. Eligible healthy participants are admitted on D-1 and receive a single oral dose of ACC017 tablets on the day of administration of each cycle under the fasting or postprandial condition, with a washout period of 7 days during the two-week period. After completing the second cycle of drug washout, participants are evaluated by the investigator and enter into the DDI study and receive a single oral dose of ACC017 tablets with FTC/TAF tablets under fasting condition.

The study is divided into screening period (no more than 28 days, D-28 to D-1), FE first cycle (D1), washout period A (D2 to D7), FE second cycle (D8), washout period B (D9 to D14), DDI period (D15), wahout period C (D16 to D21), and discharge (D22) visits.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteering to sign the informed consent and able to follow protocol-defined procedural requirements;
2. Aged 18 to 55 years (inclusive);
3. Male weighing ≥ 50.0 kg, female weighing ≥ 45.0 kg, and body mass index (BMI) = weight(kg)/height^2 (m^2) within the range of 18.5~26 kg/m^2 (inclusive);
4. Women of child-bearing potential (WOCBP) or men without a birth plan (including sperm or egg donation) and agreeing to use effective contraception (including one or more non-pharmacological contraceptives or non-heterosexual sexual activity in daily life) from 1 month prior to informed consent up to 3 months after the last dose of the study medication;
5. No history of significant medical or surgical illness, and normal results on vital signs, physical examination, 12-lead electrocardiogram (ECG), laboratory tests, chest X-ray and abdominal ultrasound examination during the screening period, or minor deviations from normal reference values that are not clinically significant in the judgment of the investigator.

Exclusion Criteria:

1. Occurrence or persistence of clinically significant abnormal conditions, including but not limited to cardiovascular, respiratory, gastrointestinal (any history of gastrointestinal disorders affecting the absorption of medications), urinary, hematologic and lymphatic, endocrine, musculoskeletal, immune, and neuropsychiatric disorders;
2. Possible or definite allergic reaction to the study drug, placebo, or any of the excipients contained, as judged by the investigator, or allergy (multiple drug and food sensitivities), or a history of allergic disease (e.g., asthma, urticaria, and eczematous dermatitis, etc.);
3. Acute illness, such as respiratory tract infections requiring antibiotic treatment, occurring from screening until study drug administration;
4. Inability to tolerate venipuncture, or history of needle-sickness or blood-sickness, or blood donation including component blood or significant blood loss (≥400 mL) or receipt of blood transfusion within 3 months prior to screening, or planning to donate blood during the trial period;
5. Dysphagia, or surgery within 6 months prior to screening, or surgery planned during the trial, or surgery that interferes with the absorption, distribution, metabolism, or excretion of the medication;
6. Smoking an average of >5 cigarettes per day within 3 months prior to screening, or inability to stop using any tobacco-based product during the trial period;
7. Average weekly alcohol consumption greater than 14 units (1 unit of alcohol ≈ 360 mL of beer, or 45 mL of 40% (alcohol by volume) spirits, or 150 mL of wine) within 3 months prior to screening or inability to discontinue use of any alcohol-containing product during the trial period, or with a positive breath test for alcohol at screening;
8. Excessive consumption of tea, coffee, and/or caffeinated beverages (more than 8 cups on average per day, 1 cup ≈ 250 mL) within 3 months prior to screening, or inability to stop consuming tea, coffee, and/or caffeinated beverages during the trial period;
9. Consumption or drinking of dragon fruit, mango, grapefruit, popcorn, or foods or beverages prepared from the aforementioned fruits, or foods or beverages containing xanthines, caffeine, or alcohol (including chocolate, tea, coffee, cola, and cocoa), or any other special diet that interferes with the absorption, distribution, metabolism, or excretion of the drug, within 48 hours prior to administration of the study medication;
10. With special dietary requirements, or cannot accept a uniform diet；
11. Use of strong or moderate CYP3A inhibitors (e.g., clarithromycin, telithromycin, ketoconazole, itraconazole and nefazodone, etc.) or strong CYP3A4 inducers (e.g., rifampicin, efavirenz, carbamazepine, phenobarbital, phenytoin, pioglitazone, St. John's wort, and glucocorticoids, etc.) within 28 days or 5 half-lives (whichever is longer) before screening；
12. Use of strong or moderate UGT1A inhibitors (e.g., silybin, ritonavir, atazanavir, quinidine, diclofenac, mycophenolic acid, and osimertinib, etc.) or strong UGT1A1 inducers (e.g., rifampicin, carbamazepine, phenobarbital, and phenytoin, etc.) within 28 days or 5 drug half-lives (whichever is longer) before screening;
13. Use of any prescription drugs, over-the-counter drugs or Chinese (herbal) medicines within 14 days or 5 drug half-lives (whichever is longer) prior to screening；
14. Vaccination (e.g., SARS-CoV-2 virus vaccine, and hepatitis B virus vaccine, etc.) within 1 month before screening, and are not suitable for enrollment as assessed by the investigator；
15. Positive for hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV) antibody, or human immunodeficiency virus (HIV) antibody, or Tponema pallidum (Tp) antibody at screening；
16. History of substance abuse within 5 years prior to screening, or positive urine drug screen at screening；
17. Females who are pregnant or lactating at the time of screening, or have a positive blood pregnancy test (for WOCBP only)；
18. Participation in any interventional clinical trials, including drugs, vaccines, or devices, etc., within 3 months prior to screening,；
19. It is not suitable for a participant to participate in this trial in the judgment of the investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-01-24 (Actual); Primary Completion 2024-04-23 (Estimated); Study Completion 2024-04-23 (Estimated)

PRIMARY OUTCOMES:
Frequency, causality, severity, and expectedness of adverse events (AEs) | Day 1 through Day 8 of Stage 1; Day 1 through Day 8 and Day 15 through Day 22 of Stage 2
  Includes Adverse Drug Reactions [ADRs], Grade 3 and above AEs, and Serious Adverse Events [SAEs], Serious Adverse Drug Reactions [SADRs], AEs resulting in treatment interruptions, AEs resulting in early withdrawal from the trial, and AEs of Special Interest [AESI]
ACC017 PK parameter: Cmax (after a single mono-drug administration under the fasting condition) | Day 1 through Day 8 of Stage 1
  Cmax is defined as the maximum observed concentration of drug
ACC017 PK parameter: C24h (after a single mono-drug administration under the fasting condition) | Day 1 through Day 8 of Stage 1
  C24h is defined as the plasma drug concentrations sampled 24 hours-post dose (C24h)
ACC017 PK parameter: AUC0-t (after a single mono-drug administration under the fasting condition) | Day 1 through Day 8 of Stage 1
  AUC0-t is defined as area under the plasma concentration-time curve from time zero to the time of the last measurable plasma concentration
ACC017 PK parameter: AUC0-∞ (after a single mono-drug administration under the fasting condition) | Day 1 through Day 8 of Stage 1
  AUC0-∞ is defined as AUC from time zero to infinity
ACC017 PK parameter: Tmax (after a single mono-drug administration under the fasting condition) | Day 1 through Day 8 of Stage 1
  Tmax is defined as the time to reach Cmax
ACC017 PK parameter: t1/2 (after a single mono-drug administration under the fasting condition) | Day 1 through Day 8 of Stage 1
  Half-life
ACC017 PK parameter: Vz/F (after a single mono-drug administration under the fasting condition) | Day 1 through Day 8 of Stage 1
  Apparent volume of distribution during terminal phase after oral administration
ACC017 PK parameter: CL/F (after a single mono-drug administration under the fasting condition) | Day 1 through Day 8 of Stage 1
  Apparent total plasma clearance of drug after oral administration
ACC017 PK parameter: λz (after a single mono-drug administration under the fasting condition) | Day 1 through Day 8 of Stage 1
  Terminal elimination rate constant
ACC017 PK parameter: AUC_%Extrap (after a single mono-drug administration under the fasting condition) | Day 1 through Day 8 of Stage 1
  Percentage of AUCinf due to extrapolation from Tlast to infinity
ACC017 PK parameter: MRT0-t (after a single mono-drug administration under the fasting condition) | Day 1 through Day 8 of Stage 1
  MRT0-t is defined as the mean retention time from time zero to the time of the last measurable plasma concentration
ACC017 PK parameter: MRT0-∞ (after a single mono-drug administration under the fasting condition) | Day 1 through Day 8 of Stage 1
  MRT0-∞ is defined as MRT from time zero to infinity

SECONDARY OUTCOMES:
Vital signs: temperature | Baseline and Day 1 through Day 8 of Stage 1; Day 1 through Day 8 and Day 15 through Day 22 of Stage 2
  Temperature in degree Celsius
Vital sign: pulse | Baseline and Day 1 through Day 8 of Stage 1; Day 1 through Day 8 and Day 15 through Day 22 of Stage 2
  Pulse in beat per minute
Vital signs: blood pressure | Baseline and Day 1 through Day 8 of Stage 1; Day 1 through Day 8 and Day 15 through Day 22 of Stage 2
  Systolic and diastolic blood pressure in millimeters (mm) of mercury (Hg)
Vital signs: respiration | Baseline and Day 1 through Day 8 of Stage 1; Day 1 through Day 8 and Day 15 through Day 22 of Stage 2
  Respiratory rate in breaths per minute
Electrocardiogram (ECG): heart rate | Baseline and Day 1 through Day 8 of Stage 1; Day 1 through Day 8 and Day 15 through Day 22 of Stage 2
  Heart rate in beat per minute
Electrocardiogram (ECG): PR interval | Baseline and Day 1 through Day 8 of Stage 1; Day 1 through Day 8 and Day 15 through Day 22 of Stage 2
  Changes in PR interval
Electrocardiogram (ECG): QRS duration | Baseline and Day 1 through Day 8 of Stage 1; Day 1 through Day 8 and Day 15 through Day 22 of Stage 2
  Changes in QRS duration
Electrocardiogram (ECG): QTc interval | Baseline and Day 1 through Day 8 of Stage 1; Day 1 through Day 8 and Day 15 through Day 22 of Stage 2
  Changes in QTc interval
ACC017 PK parameter: Cmax | Day 1 through Day 8 and Day 15 through Day 22 of Stage 2
  ACC017 Cmax after single postprandial single-drug administration，ACC017 Cmax after a single coadministration under the fasting condition and FTC and TAF Cmax after a single coadministration under the fasting condition
ACC017 PK parameter: C24h | Day 1 through Day 8 and Day 15 through Day 22 of Stage 2
  ACC017 C24h after single postprandial single-drug administration，ACC017 C24h after a single coadministration under the fasting condition and FTC and TAF C24h after a single coadministration under the fasting condition
ACC017 PK parameter: AUC0-t | Day 1 through Day 8 and Day 15 through Day 22 of Stage 2
  ACC017 AUC0-t after single postprandial single-drug administration，ACC017 AUC0-t after a single coadministration under the fasting condition and FTC and TAF AUC0-t after a single coadministration under the fasting condition
ACC017 PK parameter: AUC0-∞ | Day 1 through Day 8 and Day 15 through Day 22 of Stage 2
  ACC017 AUC0-∞ after single postprandial single-drug administration，ACC017 AUC0-∞ after a single coadministration under the fasting condition and FTC and TAF AUC0-∞ after a single coadministration under the fasting condition
ACC017 PK parameter: Tmax | Day 1 through Day 8 and Day 15 through Day 22 of Stage 2
  ACC017 Tmax after single postprandial single-drug administration，ACC017 Tmax after a single coadministration under the fasting condition and FTC and TAF Tmax after a single coadministration under the fasting condition
ACC017 PK parameter: t1/2 | Day 1 through Day 8 and Day 15 through Day 22 of Stage 2
  ACC017 t1/2 after single postprandial single-drug administration，ACC017 t1/2 after a single coadministration under the fasting condition and FTC and TAF t1/2 after a single coadministration under the fasting condition
ACC017 PK parameter: Vz/F | Day 1 through Day 8 and Day 15 through Day 22 of Stage 2
  ACC017 Vz/F after single postprandial single-drug administration，ACC017 Vz/F after a single coadministration under the fasting condition and FTC and TAF Vz/F after a single coadministration under the fasting condition
ACC017 PK parameter: CL/F | Day 1 through Day 8 and Day 15 through Day 22 of Stage 2
  ACC017 CL/F after single postprandial single-drug administration，ACC017 CL/F after a single coadministration under the fasting condition and FTC and TAF CL/F after a single coadministration under the fasting condition
ACC017 PK parameter: λz | Day 1 through Day 8 and Day 15 through Day 22 of Stage 2
  ACC017 λz after single postprandial single-drug administration，ACC017 λz after a single coadministration under the fasting condition and FTC and TAF λz after a single coadministration under the fasting condition
ACC017 PK parameter: AUC_%Extrap | Day 1 through Day 8 and Day 15 through Day 22 of Stage 2
  ACC017 AUC_%Extrap after single postprandial single-drug administration，ACC017 AUC_%Extrap after a single coadministration under the fasting condition and FTC and TAF AUC_%Extrap after a single coadministration under the fasting condition
ACC017 PK parameter: MRT0-t | Day 1 through Day 8 and Day 15 through Day 22 of Stage 2
  ACC017 MRT0-t after single postprandial single-drug administration，ACC017 MRT0-t after a single coadministration under the fasting condition and FTC and TAF MRT0-t after a single coadministration under the fasting condition
ACC017 PK parameter: MRT0-∞ | Day 1 through Day 8 and Day 15 through Day 22 of Stage 2
  ACC017 MRT0-∞ after single postprandial single-drug administration，ACC017 MRT0-∞ after a single coadministration under the fasting condition and FTC and TAF MRT0-∞ after a single coadministration under the fasting condition

CONTACTS AND LOCATIONS:
Overall Officials: Fujie Zhang, M.D., Ph.D., Principal Investigator — Beijing Ditan Hospital; Chaoying Hu, Ph.D., Principal Investigator — Beijing Ditan Hospital
Locations (1):
- Beijing Ditan Hospital Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No